CLINICAL TRIAL: NCT04722952
Title: an Single Center，Single Arm, Phase 3 Study to Evaluate Efficacy and Safety of PD-1 Inhibitor Combined With Azacytidine and HAG Regimen for Patients With Relapsed or Refractory Acute Myeloid Leukemia.
Brief Title: PD-1 Inhibitor Combined With Azacytidine and Homoharringtonine，Cytarabine, G-CSF for Refractory or Relapsed AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2020
Record Dates: First submitted 2020-12-21; First posted 2021-01-25 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Immunotherapy; Refractory Leukemia; Relapsed Adult AML; Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Refractory or Relapsed; Azacytidine; HAG regimen; PD-1 inhibitor
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Recurrence | interventions — visilizumab; Azacitidine; Homoharringtonine; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-PD-1 mAb Combined With Azacytidine and HAG regimen (Experimental): Anti-PD-1 mAb combined with DNA methyltransferase inhibitor Azacytidine and HAG regimen
  Interventions: Drug: Visilizumab

INTERVENTIONS:
Drug: Visilizumab — Azacytidine 75mg/(m2.d) by IV on days 1-7 of every cycle. Anti-PD-1 mAb 200mg by IV on day 8 of every cycle. Homoharringtonine(HHT) 2mg/(m2.d) by IV on days 1-6 of every cycle Cytarabine 10mg/(m2.d) by SC on days 1-7 of every cycle Granulocyte colony-stimulating factor(G-CSF) 300ug/d by SC on days 1-7 of every cycle，until absolute neutrophil count(ANC) > 5X109／L or white blood cell（WBC）> 20X109／L.
  Other Names: Azacytidine; Homoharringtonine; Cytarabine

SUMMARY:
This is an single center, single arm, phase 3 study to evaluate efficacy and safety of PD-1 Inhibitor combined with DNA methyltransferase inhibitor Azacytidine and HAG regimen for patients with relapsed and refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Treatment for Acute Myeloid Leukemia（AML） that has not responded to treatment (refractory) or has returned after treatment (relapsed) often do not work. Researchers want to see if an immunotherapy drug, combined with a less intense chemotherapy, may be able to help.

ELIGIBILITY:
Inclusion Criteria:

* Chinese guidelines for the diagnosis and treatment of relapsed and refractory acute myeloid leukemia (2017 edition)，excludes acute promyelocytic leukemia (M3、APL)

  * Hematopoietic stem cell transplantation ≥3 months, Discontinue immunosuppressant ≥3 weeks, Patients without graft-versus-host disease；
  * Be at least 18 years of age on day of signing informed consent.
  * Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group（ECOG） Performance Scale
  * Demonstrate adequate organ function as defined below, all screening labs should be performed before treatment initiation：

    1. ALT(SGPT) less than or equal to 2.5 × Upper Limit of Norma（ULN）；
    2. AST (SGOT) less than or equal to 2.5 × ULN；
    3. Serum total bilirubin Less than or equal to 2.0 × ULN Note: If total bilirubin >2.0×ULN, subjects with Gilbert syndrome records are allowed to join the group
    4. Serum Creatinine ≥ 30 mL/min
    5. Total white blood cell (WBC) count ≤10,000/µL； Note: hydroxyurea therapy is allowed to reduce white blood cells to meet this inclusion criteria.white blood cells should be determined ≥24 hours after the last hydroxyurea administration. Final hydroxyurea administration should not ≤3 days prior to the first azacytidine administration.
  * Treatment without anthracycline or demethylation. Ability to comprehend the investigational nature of the study and provide informed consent

Exclusion Criteria:

* Patients with chronic myeloid leukemia，AML of other myeloproliferative disorders Malignant neoplasms with other progression Those who can not control severe infections and other underlying diseases can not tolerate chemotherapy Patients with cardiac insufficiency： ejection fraction (EF)<30%，New York Heart Association（NYHA） standards，Cardiac insufficiency II or above Patients with liver and kidney dysfunction：Serum bilirubin (SB)≥2mg/dl，AST is 2.5 times higher than normal upper limit, serum creatinine (SCr) is more than 2.5 mg/dl Serious mental illness uncooperative Refusal to join the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission， Incomplete blood count recovery，Partial remission（CR+CRi+PR） | 8 months
  Number of Participants (Responders) Achieving CR+CRi+PR After the Eighth Cycle Treatments

SECONDARY OUTCOMES:
Overall Response Rate （ORR） | 8 months
  Number of Participants (Responders) Achieving Overall Response Rate(ORR) After the Eighth Cycle Treatments
Overall survival (OS) | 3 years
  time from randomization to death from any cause
Event free survival（EFS） | 3 years
  The time between the beginning of the group and the occurrence of any event, including death, progression of the disease, chemotherapy regimen, conversion to chemotherapy, addition of other treatment, occurrence of fatal or intolerable side effects, etc
Progression free survival（PFS） | 3 years
  Time between the beginning of randomization and the progression (in any way) of tumorigenesis or (for any reason) death

CONTACTS AND LOCATIONS:
Overall Officials: Han Yue, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thol F, Schlenk RF, Heuser M, Ganser A. How I treat refractory and early relapsed acute myeloid leukemia. Blood. 2015 Jul 16;126(3):319-27. doi: 10.1182/blood-2014-10-551911. Epub 2015 Apr 7. PMID 25852056
- [Background] Price SL, Lancet JE, George TJ, Wetzstein GA, List AF, Ho VQ, Fernandez HF, Pinilla-Ibarz J, Kharfan-Dabaja MA, Komrokji RS. Salvage chemotherapy regimens for acute myeloid leukemia: Is one better? Efficacy comparison between CLAG and MEC regimens. Leuk Res. 2011 Mar;35(3):301-4. doi: 10.1016/j.leukres.2010.09.002. Epub 2010 Nov 24. PMID 21109304
- [Background] Tallman MS, Wang ES, Altman JK, Appelbaum FR, Bhatt VR, Bixby D, Coutre SE, De Lima M, Fathi AT, Fiorella M, Foran JM, Hall AC, Jacoby M, Lancet J, LeBlanc TW, Mannis G, Marcucci G, Martin MG, Mims A, O'Donnell MR, Olin R, Peker D, Perl A, Pollyea DA, Pratz K, Prebet T, Ravandi F, Shami PJ, Stone RM, Strickland SA, Wieduwilt M, Gregory KM; OCN; Hammond L, Ogba N. Acute Myeloid Leukemia, Version 3.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 Jun 1;17(6):721-749. doi: 10.6004/jnccn.2019.0028. PMID 31200351
- [Background] Christman JK. 5-Azacytidine and 5-aza-2'-deoxycytidine as inhibitors of DNA methylation: mechanistic studies and their implications for cancer therapy. Oncogene. 2002 Aug 12;21(35):5483-95. doi: 10.1038/sj.onc.1205699. PMID 12154409
- [Background] Keating GM. Azacitidine: a review of its use in higher-risk myelodysplastic syndromes/acute myeloid leukaemia. Drugs. 2009;69(17):2501-18. doi: 10.2165/11202840-000000000-00000. PMID 19911860
- [Background] Gao S, Li Z, Fu JH, Hu XH, Xu Y, Jin ZM, Tang XW, Han Y, Chen SN, Sun AN, Wu DP, Qiu HY. Decitabine in the Treatment of Acute Myeloid Leukemia and Myelodysplastic Syndromes, Which Combined with Complex Karyotype Respectively. Asian Pac J Cancer Prev. 2015;16(15):6627-32. doi: 10.7314/apjcp.2015.16.15.6627. PMID 26434886
- [Background] Orskov AD, Treppendahl MB, Skovbo A, Holm MS, Friis LS, Hokland M, Gronbaek K. Hypomethylation and up-regulation of PD-1 in T cells by azacytidine in MDS/AML patients: A rationale for combined targeting of PD-1 and DNA methylation. Oncotarget. 2015 Apr 20;6(11):9612-26. doi: 10.18632/oncotarget.3324. PMID 25823822
- [Background] Daver N, Garcia-Manero G, Basu S, Boddu PC, Alfayez M, Cortes JE, Konopleva M, Ravandi-Kashani F, Jabbour E, Kadia T, Nogueras-Gonzalez GM, Ning J, Pemmaraju N, DiNardo CD, Andreeff M, Pierce SA, Gordon T, Kornblau SM, Flores W, Alhamal Z, Bueso-Ramos C, Jorgensen JL, Patel KP, Blando J, Allison JP, Sharma P, Kantarjian H. Efficacy, Safety, and Biomarkers of Response to Azacitidine and Nivolumab in Relapsed/Refractory Acute Myeloid Leukemia: A Nonrandomized, Open-Label, Phase II Study. Cancer Discov. 2019 Mar;9(3):370-383. doi: 10.1158/2159-8290.CD-18-0774. Epub 2018 Nov 8. PMID 30409776
- [Background] Ivanoff S, Gruson B, Chantepie SP, Lemasle E, Merlusca L, Harrivel V, Charbonnier A, Votte P, Royer B, Marolleau JP. 5-Azacytidine treatment for relapsed or refractory acute myeloid leukemia after intensive chemotherapy. Am J Hematol. 2013 Jul;88(7):601-5. doi: 10.1002/ajh.23464. Epub 2013 May 30. PMID 23619977
- [Background] Itzykson R, Thepot S, Berthon C, Delaunay J, Bouscary D, Cluzeau T, Turlure P, Prebet T, Dartigeas C, Marolleau JP, Recher C, Plantier I, Stamatoullas A, Devidas A, Taksin AL, Guieze R, Caillot D, Vey N, Ades L, Ifrah N, Dombret H, Fenaux P, Gardin C. Azacitidine for the treatment of relapsed and refractory AML in older patients. Leuk Res. 2015 Feb;39(2):124-30. doi: 10.1016/j.leukres.2014.11.009. Epub 2014 Nov 24. PMID 25524177
- [Background] Santini V, Ossenkoppele GJ. Hypomethylating agents in the treatment of acute myeloid leukemia: A guide to optimal use. Crit Rev Oncol Hematol. 2019 Aug;140:1-7. doi: 10.1016/j.critrevonc.2019.05.013. Epub 2019 May 25. PMID 31153036

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT04722952/Prot_SAP_ICF_000.pdf